CLINICAL TRIAL: NCT00630838
Title: Probiotic Prophylaxis of Hirschprung's Disease Associated Enterocolitis (HAEC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Daniel H. Teitelbaum, Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VSL-N007177
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-04

CONDITIONS: Hirschsprung Disease
Keywords: Hirschsprung disease; enterocolitis; probiotics
MeSH Terms: conditions — Hirschsprung Disease; Enterocolitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): VSL#3 probiotic
  Interventions: Drug: VSL#3
- 2 (Placebo Comparator): Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (4 sachets) of placebo will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (2 sachets) daily in the same amount of formula or breast milk Initiation: within one week of pullthrough Duration: 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSL#3 — Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (360 billion bacteria or 4 sachets) of VSL#3 will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (180 billion bacteria or 2 sachets) daily in the same amount of formula or breast milk.
  E.2.6. Time of start of probiotics: Probiotic vs. placebo will begin once the infant has reached full oral feeding.
  Arms: 1
Drug: Placebo — Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (4 sachets) of placebo will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (2 sachets) daily in the same amount of formula or breast milk Initiation: within one week of pullthrough Duration: 3 months
  Arms: 2

SUMMARY:
Prospective, randomized, controlled trial to test if post-operative administration of probiotics in HD patients will lead to a reduction in the occurrence of HAEC.

DETAILED DESCRIPTION:
To test the hypothesis that probiotics will decrease the risk of post pull-through enterocolitis by randomizing patients to receive either probiotics or placebo for the first 3 months after surgical treatment for HD.

E.1. Design: This study will be a prospectively performed, multi-center, double blinded, study drug versus placebo controlled study. It will test the hypothesis that post-operative administration of probiotics in HD patients will lead to a reduction in the occurrence of HAEC E.2. Study medication: VSL#3 (VSL Pharmaceuticals, Inc., Ft. Lauderdale, FL) was provided in packets, each of which contained 900 billion viable lyophilized bacteria of 4 strains of Lactobacillus (L. casei, L. plantarum, L. acidophilus, and L. delbrueckii subsp. bulgaricus), 3 strains of Bifidobacterium (B. longum, L. breve, and B. infantis), and 1 strain of Streptococcus salivarius subsp. thermophilus (designated hereafter as S. thermophilus). Maize starch was included as filler. Placebo was provided in identical bags containing 3 g of maize starch. VSL#3 and placebo were administered once each night. The taste and smell of the active drugs were not readily identifiable.

E.2.1. Formulation of the study drug: The drug will be delivered to patient's families in individual packets. The families will be instructed to administer the probiotic as appropriately diluted in 2 ounces of either expressed human milk or formula.

E.2.2. FDA approval number: VSL#3 is now a "medical food" in the US and does not need FDA approval.

E.2.3. Medication suppliers: VSL Pharmaceuticals, Inc., Ft. Lauderdale, FL E.2.4.Funds for medication: It is anticipated that the VSL Pharmaceutical Corporation will donate sufficient drug and placebo for the completion of this study. Additional funds for IRB approval and costs of dispensing drug/placebo via the Investigational Drug Service are requested from the VSL Pharmaceutical Corporation.

E.2.5. Dosing and frequency: Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (360 billion bacteria or 4 sachets) of VSL#3 will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (180 billion bacteria or 2 sachets) daily in the same amount of formula or breast milk.

E.2.6. Time of start of probiotics: Probiotic vs. placebo will begin once the infant has reached full oral feeding.

E.2.7. Duration of the study: Upon initiation of probiotics vs. placebo administration, administration will continue for 3 months. Follow up will continue for an additional 3 month period after termination of probiotic administration.

E.3. Study population: Study candidates will include all infants (newborn to 1 year of age) who undergo a definitive pullthrough for Hirschsprung disease.

E.3.1. Study Sites: This study will be conducted in four large pediatric surgery centers including:

* C.S. Mott Children's Hospital, Ann Arbor, Michigan, USA
* Children's Hospital of Buffalo, Buffalo, New York, USA
* Hospital for Sick Kids, Toronto, Ontario, Canada
* Tanta University, Tanta, Egypt

And the study will include all pediatric patients diagnosed to have HD and will be subjected to definitive pullthrough procedure. Each of these sites contains a quaternary level of pediatric surgical care, and treats a large number of patients with HD on a yearly basis. The key advantage of Tanta University is that this Hospital group treats three-fold more HD patients on a yearly basis than the other Sites, and has a very highly motivated staff with research interests in HAEC.

E.3.2. Method of Patient Recruitment: The study coordinator, co-investigator and collaborator at each site will conduct study orientations for the neonatal staff which will include staff physicians, training-fellows, house officers and nurses who work in the unit. These orientations will help alert the staff as to who are potential candidates for the study. In addition, the study coordinator will check each day for new admissions to the neonatal intensive care unit for potential candidates. It will be the study coordinator's responsibility to consent the parent/guardian and write orders for the study. No preference for a specific sex, race or ethnic background will be given.

E.3.3. Randomization: the study will be double blinded study and the randomization will be conducted by the hospital pharmacist whom will be responsible of dispensing the medication to the patients after coding it with a special code related to the patient ID and the records is kept with the pharmacist till the end of the study. Physicians and other caregivers will be blinded as to who is receiving placebo or study drug. Only the pharmacist at the Investigational Drug Service (or similar service) will be aware of the assignment. Each patient will receive a study number which will identify the patient. The number will allow for confidentiality while simultaneously allowing patient identification by the principal investigator at each center if it should it be necessary.

E.3.4.Mechanisms of drug / placebo distribution: The anticipated number of patients to be enrolled in this study in each participating center has been calculated according to previous records of the center. According to this number, the drug/placebo distribution will be done. The responsible group for the blindness of the study and distribution of the drug will be the pharmacist in each center and he/she will keep codes for each patient not to be broken except at the end of the study. The pharmacist is also responsible for dispensing the drug and placebo packets to the patients as monthly supplies and should inform the patient guardian to bring the empty packs before receiving the new medication to ensure compliance of the patients to the study.

E.3.5. Removal from protocol after enrollment: Although all patients will be treated as intent to treat, physicians may remove infants from the protocol for a number of reasons: First, if parent or guardian requests study withdrawal, and this will be honored. Second, if it is the opinion of the caring physician that participation in the study protocol may lead to undo harm of the child.

E.3.6. Guidelines for uniformity of patient care: As these studies will be performed at a multiple sites, a series of guidelines will need to be followed by each site. Prior to the initiation of the study, investigators and their study monitor will meet and discuss enrollment criteria, case report forms (CRF, see Appendix I) and review protocols for the performance of probiotics administration and monitoring of infants. The treatment specifications listed above will serve as an outline for definitive guidelines. Finally, a firm agreement on the definition of HAEC will be established.

E.3.7. Monitoring: Each site will specify a study monitor who will be responsible for data collection and monitoring infants for protocol compliance and the development of adverse events (AEs, see Appendix II). The study monitor will be responsible for data transmission for data collection and analysis. He/she will also be responsible for informing the Investigator and the respective IRBs of adverse events. When there is an adverse event which is believed to have a relation to the performance of this study or a significant adverse event (SAE), they will be responsible for reporting this within 48 hours to both their IRB, and all other investigators. In a similar time, a report to the FDA will be done. Yearly reporting of all AEs to each IRB and the FDA will be done.

E.3.8. Safety and Regulatory Issues: Full IRB approval from each participating institution will be attained, and IRB will be apprised of the multi-center design as well as names of other participating sites.

E.3.9. Data Obtained:

E.4.0. Primary Outcome Measure: The primary outcome measure will be the diagnosis of Hirschsprung-associated enterocolitis (HAEC).

The severity of clinical episodes of HAEC will be stratified into three grades according to established clinical grading system as follows (11):

Grade I: mild explosive diarrhea, mild to moderate abdominal distension, no significant systemic manifestations (fever, anorexia, weight loss, tachycardia).

Grade II: moderate explosive diarrhea, moderate to sever abdominal distension associated with mild to moderate systemic manifestations.

Grade III: explosive diarrhea, marked abdominal distension, shock, or impending shock.

E.4.1. Secondary Outcome Measures: Secondary outcome measures will be to measure the expression of MUC-2 and MUC-3 expressed proteins in the stools of study patients.

Mucins will be detected by using a modified Western immunoblot technique of stool specimens as previously described.

Finally, we will attempt to correlate if there are additional clinical benefits of probiotics in HD, by examining the number of un-scheduled clinic visits or emergency visits, the stooling pattern, and the growth curve in probiotic treated group versus the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for enrollment will include all pediatric patients suffering from HD at an age of 12 months or younger. All patients will require consent by either parent or adult guardian

Exclusion Criteria:

* Patients will be excluded if children that are deemed hemodynamically unstable and require immediate operative intervention, age more than one year of age, as this may mean very delay in diagnosis and may affect the study results, or infants having major congenital anomalies with short life expectancy. Additional exclusion criteria are those patients' parents or adult guardian who refuse to undergo randomization. Finally, those children who are transferred to another non-participating hospital will be excluded.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Teitelbaum, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Buffalo, Buffalo, New York

REFERENCES:
- [Derived] El-Sawaf M, Siddiqui S, Mahmoud M, Drongowski R, Teitelbaum DH. Probiotic prophylaxis after pullthrough for Hirschsprung disease to reduce incidence of enterocolitis: a prospective, randomized, double-blind, placebo-controlled, multicenter trial. J Pediatr Surg. 2013 Jan;48(1):111-7. doi: 10.1016/j.jpedsurg.2012.10.028. PMID 23331802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants scheduled for endorectal pullthrough who were consented were randomized, but 1 died following the surgery prior to any study specific placebo usage.
Groups:
- VSL#3 Probiotic: VSL#3 probiotic
  VSL#3 : Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (360 billion bacteria or 4 sachets) of VSL#3 will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (180 billion bacteria or 2 sachets) daily in the same amount of formula or breast milk.
  E.2.6. Time of start of probiotics: Probiotic vs. placebo will begin once the infant has reached full oral feeding.
- Placebo: Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (4 sachets) of placebo will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (2 sachets) daily in the same amount of formula or breast milk Initiation: within one week of pullthrough Duration: 3 months
  Placebo : Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (4 sachets) of placebo will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (2 sachets) daily in the same amount of formula or breast milk Initiation: within one week of pullthrough Duration: 3 months
Period: Overall Study
Arm/Group | VSL#3 Probiotic | Placebo
Started | 32 | 30
Completed | 32 | 28
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VSL#3 Probiotic | Placebo | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 32 (7.6) | 28 (4.9) | 30 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 18 | 25 | 43
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
  Egypt | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Diagnosed With Hirschsprung-associated Enterocolitis (HAEC).
Description: The primary outcome measure is reporting the number of participants diagnosed with Hirschsprung-associated enterocolitis (HAEC) after pullthrough procedure.
Time Frame: 6 months post-pullthrough
Measure: Number; unit: participants
Groups:
- VSL#3 Probiotic: VSL#3: Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (360 billion bacteria or 4 sachets) of VSL#3 will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (180 billion bacteria or 2 sachets) daily in the same amount of formula or breast milk.
  E.2.6. Time of start of probiotics: Probiotic vs. placebo will begin once the infant has reached full oral feeding.
Arm/Group | VSL#3 Probiotic | Placebo
Number analyzed (Participants) | 32 | 28
participants | 10 | 7
Statistical Analysis 1: Comparison: VSL#3 Probiotic vs Placebo; Test type: Superiority or Other; p = 0.897, t-test, 2 sided

2. Primary Outcome: Severity of Clinical Episodes of HAEC
Description: The severity of clinical episodes of HAEC will be stratified into three grades (mild, moderate, or severe). Grades of severity reported are based on first episodes.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- VSL#3 Probiotic: VSL#3 : Dosing will be based on patient weight. For those infants greater or equal to 5 kg, one gram (360 billion bacteria or 4 sachets) of VSL#3 will be administered into 3 ounces of either expressed breast milk or formula daily. For patients under 5 kg, 0.5 gm (180 billion bacteria or 2 sachets) daily in the same amount of formula or breast milk.
  E.2.6. Time of start of probiotics: Probiotic vs. placebo will begin once the infant has reached full oral feeding.
Arm/Group | VSL#3 Probiotic | Placebo
Number analyzed (Participants) | 32 | 28
participants
  HAEC Severity, Mild | 3 | 6
  HAEC Severity, Moderate | 6 | 0
  HAEC Severity, Severe | 1 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | VSL#3 Probiotic | Placebo
Serious Adverse Events (participants affected / at risk) | 10/32 | 7/28
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VSL#3 Probiotic (N=32) | Placebo (N=28)
Hirschsprung Associated Enterocolitis (HAEC) (Gastrointestinal disorders) | 10 | 7

LIMITATIONS AND CAVEATS:
The secondary outcome measure was defined before beginning the study as the measure of the expression of MUC-2 and MUC-3 expressed proteins in the stools of study patients. However, stool samples were not collected and this analysis was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No